CLINICAL TRIAL: NCT02470546
Title: Metformin Experience on Minimal Hepatic Encephalopathy in Patients With Liver Cirrhosis
Brief Title: Metformin Experience on Minimal Hepatic Encephalopathy
Acronym: EME
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EME-2015
Record Dates: First submitted 2014-09-04; First posted 2015-06-12 (Estimated); Last update posted 2015-06-12 (Estimated); Status verified 2015-06

CONDITIONS: Liver Cirrhosis; Hepatic Encephalopathy
Keywords: Hepatic encephalopathy; Metformin; Liver cirrhosis
MeSH Terms: conditions — Liver Cirrhosis; Hepatic Encephalopathy | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metformin (Active Comparator): Patients receiving metformin
  Interventions: Drug: Metformin
- Placebo (Placebo Comparator): Patients receiving placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin — Metformin 1000mg twice a day
  Other Names: Drug 1
  Arms: Metformin
Drug: Placebo — Placebo 1000mg twice a day
  Other Names: Drug 2
  Arms: Placebo

SUMMARY:
Primary aim:

-To assess the effect of metformin use on the treatment of minimal hepatic encephalopathy in patients with liver cirrhosis.

Secondary aim:

-To evaluate if metformin is a safety drug in patients showing liver cirrhosis.

DETAILED DESCRIPTION:
In this study, 30 patients will be included divided in two arms. Investigators and patients will not know the treatment used (double blind).

Arm 1: Metformin 1000mg twice a day (2000 mg/day), during 12 weeks. Arm 2: Placebo 1000mg twice a day (2000mg/day), during 12 weeks.

At the end of the study, patients will be followed-up 8 weeks more to control the appearance of adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients with > 18 years old
* Patients with the results of all the factors evaluable at the time of inclusion
* Patients who have accepted their participation in the study through informed consent
* Patients showing liver cirrhosis by ultrasound, transient elastography or liver biopsy
* Patients showing minimal hepatic encephalopathy (PHES < 4 or Critical Flicker Frequency < 39 Hz)

Exclusion Criteria:

* Patients with any contraindications to the drugs used
* Patients showing type 1 diabetes mellitus
* Patients showing type 2 diabetes mellitus and previous or current use of exogenous insulin, metformin or other oral antidiabetic drug

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-06 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with Minimal hepatic encephalopathy | 12 weeks
  Measurement of the results of critical flicker frequency after 12 weeks of metformin treatment

SECONDARY OUTCOMES:
Number of patients with Minimal hepatic encephalopathy | 12 weeks
  Measurement of the results of PHES after 12 weeks of metformin treatment

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Romero-Gomez, PhD, MD, Principal Investigator — Valme University Hospital
Locations (1):
- Fundación Pública Andaluza para la Gestión de la investigación en salud de Sevilla (FISEVI), Seville, Spain